CLINICAL TRIAL: NCT06885216
Title: Patient Characteristics, Prognosis and Outcome Measures in Patients with Concurrent Neck Associated Headache Operated for Degenerative Cervical Radiculopathy. a Population Based Study by NORspine
Brief Title: Outcomes After Surgery for Degenerative Cervical Radiculopathy in Patients with Concurrent Headache
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Tore Solberg, Consultant Neurosurgeon, University Hospital of North Norway
Other Study IDs: 03276-1
Record Dates: First submitted 2025-03-18; First posted 2025-03-20 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-04

CONDITIONS: Headache; Cervical Radiculopathy
MeSH Terms: conditions — Headache; Radiculopathy | interventions — Gene Fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Anterior cervical discectomy and fusion/ posterior decompression

SUMMARY:
Surgery for degenerative cervical radiculopathy (DCR) is one of the most common causes of neck surgery. The typical surgical indication is radicular pain (arm pain) caused by nerve impingement. However, many patients also report varying degrees of pain in the neck and head. This headache, often referred to as cervicogenic headache (CEH), is believed to result from the convergence of trigeminal afferents and the upper three cervical spinal nerves in structures such as facet joints, ligaments, cervical muscles, intervertebral and nerve roots.

The diagnostic criteria used to distinguish CEH from the other types of headaches are based on low to moderate evidence and can be challenging due to their similar clinical presentations. Nevertheless, headache disorders are a common cause of disability and many patients undergoing surgery for DCR report headache. However, prior reports assessing headache in patients surgically treated for DCR are limited by small sample sizes, inconsistent inclusion criteria and outcome measures. Consequently, there is limited understanding about the frequency of DCR associated headache and whether these patients experience meaningful improvements in their headache following surgical treatment.

The aims of this study are to assess 1) the frequency of DCR associated headache in patients operated for DCR, 2) the minimal clinical important change for NRS headache 3) if DCR associated headache is an independent prognostic factor for neck pain-related disability and 4) if patients experience improvement in their headache 12 months after surgery for DCR.

DETAILED DESCRIPTION:
Hypothesis:

Our null hypothesis is that DCR patients with and without concomitant headache have similar outcomes after surgery. Our alternative hypothesis is that concomitant headache is a negative predictor for a favourable outcome of DCR surgery, i.e. an effect size less than the MCIC value for improvement.

Data source:

The project will use prospectively collected data from the Norwegian Registry for Spine Surgery (NORspine). The NORspine is a comprehensive national clinical registry, with a capture rate of patients operated for DCR of 75% from 2021 and a response rate at 12 months follow-up of 80% in 2022. The coverage rate at the institutional level is 95-100%.

Analyses and reporting will be conducted according to the methodology proposed by PROGRESS (prognosis research strategy) framework, and reported according to the STROBE (strengthening the reporting of observational studies in epidemiology) statement.

Data collection:

Demographic variables, smoking, educational level, duration of symptoms, status on sick leave, working and disability status are collected at admission (baseline). Comorbidity, diagnosis, treatment as well as perioperative complications are recorded by surgeons. Patient reported outcome measures (PROMs) are recorded at admission (baseline) and 3- and 12 months follow-up time) after surgery.

Statistical analyses:

The invastigators will select patients with both headache and neck pain assessed with the NRS to assess the frequency of DCR associated headache.

To determine the MCIC of DCR associated headache the invastigators will use the global perceived effect (GPE) scale as the external criterion (anchor). The invastigators will assess the mean NRS headache score at 12 months, change score between baseline and 12 months follow-up and the corresponding percentage change score. A cut-off value for the NRS headache MCIC will be obtained by assessing values of sensitivity and specificity receiver operating curve (ROC).

Univariable and multivariable analyses will be used to evaluate if NRS headache is a potential prognostic factor against the NDI (35% improvement (yes/no) using binary logistic regression, adjusted for a priori selection of confounding factors. A p-value of <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion criteria:

* Patients 16 years or above and operated for degenerative cervical radiculopathy (disc herniation or spondylosis)
* Single level or multiple (primary surgery)
* Anterior cervical discectomy and fusion with or without plate
* Artificial cervical disc replacement

Exclusion criteria:

* Degenerative cervical myelopathy, tumour, inflammation, infection and trauma
* Previous surgery in the cervical spine
* Corpectomy
* Posterior approach as laminectomi with or without fusion and foramenotomi

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will include consecutive patients operated for DCR in public and private hospitals and registered in the NORspine from January 2012 to December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Neck disability index (NDI) | 3- and 12 months
  The NDI measures how neck pain affects daily life in the following domains: pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation, using a 6-point ordinal scale (0-5). The 10 items are summarized and recalculated to a percentage score ranging from 0 to 100 (no to maximum disability). The NDI percentage change will be dichotomized to 35% improvement (yes/no).

SECONDARY OUTCOMES:
NDI headache | 3- and 12 months
  NDI headache scale contains the following responses: (0) "I have no headaches at all", (1) "I have slight headaches, which come infrequently", (2) "I have moderate headaches, which come infrequently", (3) "I have moderate headaches, which come frequently", (4) "I have severe headaches, which come frequently" and (5) "I have headaches almost all the time".
Numeric rating scale for neck pain (NRS-NP) | 3- and 12 months
  NRS-NP assesses pain severity ranging from 0 to 10 ("no" to "worst conceivable pain").
Numeric rating scale for arm pain (NRS-AP) | 3- and 12 months
  NRS-AP assesses pain severity ranging from 0 to 10 ("no" to "worst conceivable pain").
NRS-HA | 3- and 12 months
  Numeric rating scale for headache (NRS-HA) assesses pain severity ranging from 0 to 10 ("no" to "worst conceivable pain").
Global perceived effect (GPE) | 3- and 12 months
  GPE scale measures the perceived benefit after surgery: (1) "completely recovered," (2) "much improved," (3) "slightly improved," (4) "unchanged," (5) "slightly worse," (6) "much worse", and (7) "worse than ever."

OTHER OUTCOMES:
EQ-5D-3L | 12 month
  EQ-5D-3L is a preference-weighted measure of health-related quality of life based on five dimensions: mobility, self-care, usual activity, pain/discomfort and anxiety/discomfort (23). The patient assesses three possible levels (3L); "none," "mild to moderate," and "severe" for each dimension. The score ranges from 0.59 to 1, where 1 corresponds to perfect health and 0 to death and negative values worse than death.

CONTACTS AND LOCATIONS:
Overall Officials: Tore Solberg, MD/PhD, Principal Investigator — University Hospital North Norway and The Arctic University of Norway

IPD SHARING:
Plan to Share IPD: No
Due to patient sensitiv data content.

REFERENCES:
- [Background] Carette S, Fehlings MG. Clinical practice. Cervical radiculopathy. N Engl J Med. 2005 Jul 28;353(4):392-9. doi: 10.1056/NEJMcp043887. No abstract available. PMID 16049211
- [Background] Bogduk N. Cervicogenic headache: anatomic basis and pathophysiologic mechanisms. Curr Pain Headache Rep. 2001 Aug;5(4):382-6. doi: 10.1007/s11916-001-0029-7. PMID 11403743
- [Background] Demont A, Lafrance S, Benaissa L, Mawet J. Cervicogenic headache, an easy diagnosis? A systematic review and meta-analysis of diagnostic studies. Musculoskelet Sci Pract. 2022 Dec;62:102640. doi: 10.1016/j.msksp.2022.102640. Epub 2022 Aug 31. PMID 36088782
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Torbjorn AF, Stolt-Nielsen A, Skaanes KO, Sjaastad O. Headache and the lower cervical spine: long-term, postoperative follow-up after decompressive neck surgery. Funct Neurol. 2003 Jan-Mar;18(1):17-28. PMID 12760410
- [Background] Liu H, Ploumis A, Wang S, Li C, Li H. Treatment of Cervicogenic Headache Concurrent With Cervical Stenosis by Anterior Cervical Decompression and Fusion. Clin Spine Surg. 2017 Oct;30(8):E1093-E1097. doi: 10.1097/BSD.0000000000000291. PMID 28937465
- [Background] Hemingway H, Riley RD, Altman DG. Ten steps towards improving prognosis research. BMJ. 2009 Dec 30;339:b4184. doi: 10.1136/bmj.b4184. No abstract available. PMID 20042483
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Background] Vernon H. The Neck Disability Index: state-of-the-art, 1991-2008. J Manipulative Physiol Ther. 2008 Sep;31(7):491-502. doi: 10.1016/j.jmpt.2008.08.006. PMID 18803999
- [Background] Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108. doi: 10.1097/00005650-199711000-00002. PMID 9366889
- [Background] Haefeli M, Elfering A. Pain assessment. Eur Spine J. 2006 Jan;15 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s00586-005-1044-x. Epub 2005 Dec 1. PMID 16320034